CLINICAL TRIAL: NCT05727475
Title: Change in Oral Health-Related Quality of Life Following Minimally Invasive Aesthetic Treatment of Anterior Teeth in Children With Molar Incisor Hypomineralization: A Prospective Clinical Study.
Brief Title: Change in OHRQOL Following Minimally Invasive Treatment of Anterior Teeth in Children With MIH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Collaborators: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 556-2021
Record Dates: First submitted 2023-02-05; First posted 2023-02-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Molar Incisor Hypomineralization
Keywords: Minimally invasive; Esthetic treatment; Oral health related quality of life; C-OHIP-SF19; Composite veneer
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Active Comparator): In this group, a composite facing will be placed on the anterior incisors to mask the opacity. Minimal invasive treatment will be done without drilling or removal of enamel. They will be asked to fill in the Child Oral Health Impact Profile-Short Form (C-OHIP-SF19) questionnaire pre and 1 month post treatment.
  Interventions: Procedure: Minimal invasive restorative treatment
- Control group (Active Comparator): In this group, fluoride gel application will be done for all teeth using 1.23% APF gel delivered through a foam tray. They will be asked to fill in the Child Oral Health Impact Profile-Short Form (C-OHIP-SF19) questionnaire pre and 1 month post treatment.
  After filling the C-OHIP-SF19 questionnaire 1 month post treatment, if the child is not happy with the appearance after fluoride gel application, a composite facing will be offered.
  Interventions: Procedure: Fluoride gel application

INTERVENTIONS:
Procedure: Minimal invasive restorative treatment — Composite veneer facing without drilling or removal of enamel
  Arms: Study group
Procedure: Fluoride gel application — Fluoride gel application 1.23%
  Arms: Control group

SUMMARY:
MIH is a prevalent developmental defect which has a negative impact on children's OHRQoL, especially when incisor opacities are present. The aim of this study is to evaluate the change in OHRQoL following minimally invasive aesthetic treatment of anterior permanent teeth opacities in children with MIH using the Arabic C-OHIP-SF19 as a data collection tool.

This RCT will be conducted on children with MIH (n=156), aged 6-16 years, at the Post Graduate (PG) clinics, Jordan University of Science and Technology (Irbid). Patients will be randomly assigned in to two groups: Study group (n=78), with anterior teeth composite facing done to mask the opacity, and control group (n=78) where fluoride gel application was done. Children will be assessed by filling the COHIP-SF19 questionnaire before and one-month after the treatment to evaluate OHRQoL changes.

DETAILED DESCRIPTION:
Background: Molar Incisor Hypomineralization (MIH) is defined as a hypomineralized lesion of the enamel as a result of different causes, mainly affecting permanent first molars and frequently associated to similar lesions (that appear as opacities) on upper and/or lower permanent incisors, causing deterioration and destruction of affected teeth because the enamel is fragile, and depending on the severity, may cause teeth to be lost.

Aim: The aim of this clinical study is to evaluate the change in oral health-related quality of life following minimally invasive aesthetic treatment of anterior permanent teeth in children with molar incisor hypomineralization using the Arabic C-OHIP-SF19 as a data collection tool.

Methods: This will be a prospective clinical study which will be performed on a group of school-children with MIH at the Post Graduate (PG) clinics, Jordan University of Science and Technology (JUST), ages 6-16 years. A total of 156 children with MIH and anterior permanent teeth opacities, requesting cosmetic improvement of one or more anterior permanent teeth will be offered a composite facing. They will be asked to fill in the Child Oral Health Impact Profile-Short Form (C-OHIP-SF19) questionnaire pre and 1 month post treatment. The patients will be divided into 2 groups (78 participants per group): Group 1: Restorative group (study group); in this group, a composite facing will be placed on the anterior incisors to mask the opacity. Minimal invasive treatment will be done without drilling or removal of enamel, unless there is caries, which will be removed in this case, and Group 2: Fluoride gel group (control group); in this group, fluoride gel application will be done for all teeth using 1.23% APF gel delivered through a foam tray. In this group, if the child is not happy with the appearance after fluoride gel application, a composite facing will be offered.

Expected results: We expect that MIH patients who undergo the minimally invasive composite facing for the anterior teeth in order to reduce the visibility of enamel opacities to have a higher score on the C-OHIP-SF19 questionnaire because the esthetic treatment can have a positive impact on the children's wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Children with MIH and who have a visible enamel opacity involving at least one anterior permanent tooth;
* Children who request improvement in their anterior permanent teeth aesthetics.

Exclusion criteria:

* Children who have an acute dental symptom and require urgent treatment;
* Children who need to undergo active treatment for their hypomineralized molars during the proposed study period (e.g., extractions) or orthodontic treatment;
* Children with any dental or facial anomaly other than MIH;
* Children with compromised incisor aesthetics due to a traumatic dental injury (crown fracture), tooth surface loss, or caries;
* Children with MIH and who do not have a visible enamel opacity involving at least one anterior permanent tooth; and
* Children with poor behavior.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 156 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
OHRQoL changes | After 1 year
  Changes OHRQoL before and after the intervention and the difference between both groups (group 1 and 2).

CONTACTS AND LOCATIONS:
Overall Officials: Ola B. Al-Batayneh, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Jordan University of Science and Technology, Irbid, Jordan

REFERENCES:
- [Background] Americano GC, Jacobsen PE, Soviero VM, Haubek D. A systematic review on the association between molar incisor hypomineralization and dental caries. Int J Paediatr Dent. 2017 Jan;27(1):11-21. doi: 10.1111/ipd.12233. Epub 2016 Apr 21. PMID 27098755
- [Background] Arheiam AA, Baker SR, Ballo L, Elareibi I, Fakron S, Harris RV. The development and psychometric properties of the Arabic version of the child oral health impact profile-short form (COHIP- SF 19). Health Qual Life Outcomes. 2017 Nov 13;15(1):218. doi: 10.1186/s12955-017-0796-4. PMID 29132377
- [Background] Broder HL, Wilson-Genderson M, Sischo L. Reliability and validity testing for the Child Oral Health Impact Profile-Reduced (COHIP-SF 19). J Public Health Dent. 2012 Fall;72(4):302-12. doi: 10.1111/j.1752-7325.2012.00338.x. Epub 2012 Apr 27. PMID 22536873
- [Background] da Costa-Silva CM, Jeremias F, de Souza JF, Cordeiro Rde C, Santos-Pinto L, Zuanon AC. Molar incisor hypomineralization: prevalence, severity and clinical consequences in Brazilian children. Int J Paediatr Dent. 2010 Nov;20(6):426-34. doi: 10.1111/j.1365-263X.2010.01097.x. Epub 2010 Aug 24. PMID 20738434
- [Background] Hasmun N, Lawson J, Vettore MV, Elcock C, Zaitoun H, Rodd H. Change in Oral Health-Related Quality of Life Following Minimally Invasive Aesthetic Treatment for Children with Molar Incisor Hypomineralisation: A Prospective Study. Dent J (Basel). 2018 Nov 1;6(4):61. doi: 10.3390/dj6040061. PMID 30388743
- [Background] Hasmun N, Vettore MV, Lawson JA, Elcock C, Zaitoun H, Rodd HD. Determinants of children's oral health-related quality of life following aesthetic treatment of enamel opacities. J Dent. 2020 Jul;98:103372. doi: 10.1016/j.jdent.2020.103372. Epub 2020 May 11. PMID 32437856
- [Background] Minamidate T, Haruyama N, Takahashi I. The development, validation, and psychometric properties of the Japanese version of the Child Oral Health Impact Profile-Short Form 19 (COHIP-SF 19) for school-age children. Health Qual Life Outcomes. 2020 Jul 11;18(1):224. doi: 10.1186/s12955-020-01469-y. PMID 32653004
- [Background] Oyedele TA, Folayan MO, Adekoya-Sofowora CA, Oziegbe EO. Co-morbidities associated with molar-incisor hypomineralisation in 8 to 16 year old pupils in Ile-Ife, Nigeria. BMC Oral Health. 2015 Mar 13;15:37. doi: 10.1186/s12903-015-0017-7. PMID 25887347
- [Background] Schwendicke F, Elhennawy K, Reda S, Bekes K, Manton DJ, Krois J. Global burden of molar incisor hypomineralization. J Dent. 2018 Jan;68:10-18. doi: 10.1016/j.jdent.2017.12.002. Epub 2017 Dec 6. PMID 29221956
- [Background] Sischo L, Broder HL. Oral health-related quality of life: what, why, how, and future implications. J Dent Res. 2011 Nov;90(11):1264-70. doi: 10.1177/0022034511399918. Epub 2011 Mar 21. PMID 21422477
- [Background] Weerheijm KL, Duggal M, Mejare I, Papagiannoulis L, Koch G, Martens LC, Hallonsten AL. Judgement criteria for molar incisor hypomineralisation (MIH) in epidemiologic studies: a summary of the European meeting on MIH held in Athens, 2003. Eur J Paediatr Dent. 2003 Sep;4(3):110-3. PMID 14529329
- [Background] William V, Messer LB, Burrow MF. Molar incisor hypomineralization: review and recommendations for clinical management. Pediatr Dent. 2006 May-Jun;28(3):224-32. PMID 16805354
- [Background] Zawaideh FI, Al-Jundi SH, Al-Jaljoli MH. Molar incisor hypomineralisation: prevalence in Jordanian children and clinical characteristics. Eur Arch Paediatr Dent. 2011 Feb;12(1):31-6. doi: 10.1007/BF03262776. PMID 21299943